CLINICAL TRIAL: NCT02700659
Title: A Clinical, Non-intervention Study of the Cxbladder Urine Test for the Detection of Recurrent Urothelial Carcinoma (UC)
Brief Title: The Cxbladder Monitoring Study
Status: Completed | Type: Observational
Sponsor: Pacific Edge Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Cxb-012-EXP-013
Record Dates: First submitted 2016-01-13; First posted 2016-03-07 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified, consented participant samples of between 5mL and 15 mL of urine, stabilized in the proprietary Cxbladder liquid, will be stored at -80ºC for further urinary diagnostic assay development and improvement.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- UC monitoring patients: Patients undergoing investigative cystoscopy for the detection of urothelial carcinoma as part of a standard-of-care schedule of investigations.
  All patients will have urine samples taken and analyzed for NMP22 ELISA, NMP22 BladderChek, urine cytology and Cxbladder.
  No results for any tests under evaluation in this study are provided to the clinician for diagnostic purposes.
  Interventions: Other: Cxbladder

INTERVENTIONS:
Other: Cxbladder — Cxbladder is a non invasive UC detection test measuring five messenger RNA (mRNA) biomarkers present at elevated levels in patients presenting with urothelial carcinoma.

SUMMARY:
The aim of this trial is to determine the performance characteristics of the Cxbladder test for the detection of recurrent urothelial carcinoma (UC) in patients with a recent history of urinary tract UC, who have been treated according to standard practice and are undergoing routine investigative cystoscopy.

The gold standard for determination of clinical truth is cystoscopy, plus any follow up investigations relating to the current visit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed positive diagnosis for primary or recurrent urinary tract UC over the past 2 years.
* Patient is undergoing investigative cystoscopies for the monitoring of recurrence of UC at intervals prescribed by a clinical practitioner
* Patient is 18 years of age or older.

Exclusion Criteria:

* Prior genitourinary manipulation (cystoscopy / catheterisation / dilation) in the 14 days before urine collection, current urinary tract infection, current or known history of urinary tract inflammatory disorder, recent history of glomerulonephritis, nephrosis or other renal inflammatory disorders, recent history of pyelonephritis
* Patient has undergone total bladder cystectomy as treatment for bladder UC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited from community and referral centres. Patients were under surveillance for recurring urothelial carcinoma monitoring, and undergoing all standard of care, including investigative cystoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with bladder cancer who are correctly identified as having cancer (true positives) and no cancer (true negatives) by the Cxbladder test. | The outcome measure will be assessed by 6 months after trial completion.
  The Cxbladder test results will be compared to that of cystoscopy, which is the gold standard method for diagnosing urothelial cancer; the true positive and true negative rates will be measured, along with the false positive and false negative rates of the test. The results will be reported as sensitivity and specificity of the Cxbladder test for detecting urothelial cancer in patients with recurrent disease.
Probability that patients identified as having cancer and no cancer by the Cxbladder test truly have cancer (positive predictive value; PPV), and truly have no cancer (negative predictive value; NPV) respectively. | The outcome measure will be assessed by 6 months after trial completion.

SECONDARY OUTCOMES:
Comparison of the Cxbladder test's sensitivity, specificity, PPV and NPV with that of Cytology. | The outcome measure will be assessed by 6 months after trial completion.
  Performance characteristics (sensitivity, specificity, PPV and NPV) of the Cxbladder test for detecting recurring urothelial cancer will be compared to urine cytology, in addition to the gold standard test (cystoscopy). All comparator tests will be carried out on the same voided urine sample used for Cxbladder tests.
Comparison of the Cxbladder test's sensitivity, specificity, PPV and NPV with that of NMP22 ELISA Assay. | The outcome measure will be assessed by 6 months after trial completion.
  Performance characteristics (sensitivity, specificity, PPV and NPV) of the Cxbladder test for detecting recurring urothelial cancer will be compared to NMP22 ELISA, in addition to the gold standard test (cystoscopy). All comparator tests will be carried out on the same voided urine sample used for Cxbladder tests.
Comparison of the Cxbladder test's sensitivity, specificity, PPV and NPV with that of NMP22 BladderChek Assay. | The outcome measure will be assessed by 6 months after trial completion.
  Performance characteristics (sensitivity, specificity, PPV and NPV) of the Cxbladder test for detecting recurring urothelial cancer will be compared to NMP22 BladderChek, in addition to the gold standard test (cystoscopy). All comparator tests will be carried out on the same voided urine sample used for Cxbladder tests.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J O'Sullivan, PhD, Study Chair — Pacific Edge Limited
Locations (11):
- United States (11):
  - Urology Centers of Alabama, Homewood, Alabama
  - Urology Center of Grove Hill, One Lake Street, New Britain, Connecticut
  - Florida Urology Associates, Orlando, Florida
  - Idaho Urologic Institute, Meridian, Idaho
  - Delaware Valley Urology, LLC, New Jersey, New Jersey
  - Premier Medical Group of the Hudson Valley, Kingston, New York
  - Weill Cornell Medical College, Department of Urology, New York, New York
  - Premier Medical Group of the Hudson Valley, New York, New York
  - Premier Medical Group of the Hudson Valley, Newburgh, New York
  - Penn State Hershey Medical Center and College of Medicine, Hershey, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Lough T, Luo Q, O'Sullivan P, Chemasle C, Stotzer M, Suttie J, Darling D. Clinical Utility of Cxbladder Monitor for Patients with a History of Urothelial Carcinoma: A Physician-Patient Real-World Clinical Data Analysis. Oncol Ther. 2018 Jun;6(1):73-85. doi: 10.1007/s40487-018-0059-5. Epub 2018 Apr 19. PMID 32700139